CLINICAL TRIAL: NCT02013765
Title: An Open-label Pilot Study of the Effect of Second-line Treatment With Herceptin Monotherapy on Time to Disease Progression in Patients With Metastatic Urothelial Cancer and HER2 Overexpression
Brief Title: A Study of Herceptin (Trastuzumab) Monotherapy in Patients With Metastatic Urothelial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was terminated prematurely because of recruitment difficulties.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17599
Record Dates: First submitted 2013-12-03; First posted 2013-12-17 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Urinary Tract Cancer
MeSH Terms: conditions — Urologic Neoplasms | interventions — Trastuzumab

ARMS (1):
- Trastuzumab Monotherapy (Experimental): Participants received an initial dose of trastuzumab 4 milligrams per kilogram (mg/kg) intravenously (IV) on Day 1, followed by weekly doses of 2 mg/kg IV beginning on Day 8 and continuing for up to 37 weeks.
  Interventions: Drug: trastuzumab

INTERVENTIONS:
Drug: trastuzumab — Initial dose of 4 mg/kg i.v on Day 1, followed by weekly doses of 2 mg/kg i.v. beginning on Day 8 and continuing for up to 37 weeks.
  Other Names: Herceptin

SUMMARY:
This study will evaluate the efficacy and safety of intravenous Herceptin in patients with metastatic urothelial cancer with disease progression during platinum-based chemotherapy. The anticipated time on study treatment is until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* metastatic urothelial cancer;
* disease progression during or after 1 prior platinum-based chemotherapy;
* measurable disease;
* HER2 overexpression (IHC [2+] or [3+]).

Exclusion Criteria:

* concomitant chemotherapy or immunotherapy;
* active or uncontrolled infection;
* solely CNS metastases;
* clinically significant cardiac disease, advanced pulmonary disease or severe dyspnoea;
* co-existing malignancies diagnosed within last 5 years, except basal cell cancer or cervical cancer in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2001-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (6):
- Germany (6):
  - Aschersleben
  - Dessau
  - Fulda
  - Leipzig
  - Marburg
  - Weiden

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab Monotherapy: Participants received an initial dose of trastuzumab 4 milligrams per kilogram (mg/kg), intravenously (IV), on Day 1, followed by weekly doses of 2 mg/kg, IV, beginning on Day 8 until tumor progression, unacceptable toxicity, participant withdrawal, or termination by sponsor.
Period: Overall Study
Arm/Group | Trastuzumab Monotherapy
Started | 5
Completed | 4
Not Completed | 1
Not completed — Trial was terminated by sponsor | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) includes all participants who received study treatment.
Groups:
- Trastuzumab Monotherapy: Participants received an initial dose of trastuzumab 4 mg/kg, IV, on Day 1, followed by weekly doses of 2 mg/kg, IV, beginning on Day 8 until tumor progression, unacceptable toxicity, participant withdrawal, or termination by sponsor.
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (8.2) [60 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) - Percentage of Participants With an Event
Description: PFS was defined as the time from the first dose of study treatment to the first documentation of objective tumor progression or to death due to any cause.
Time Frame: Screening, every 3 months during treatment (up to 37 weeks), and at end of treatment
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 5
percentage of participants | 80.0

2. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: OS was defined as the time from the start of study treatment to date of death due to any cause.
Time Frame: Screening, every 4 weeks during treatment (up to 37 weeks), at end of treatment, and every 3 months thereafter
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 5
percentage of participants | 80.0

3. Secondary Outcome: Overall Survival - Time to Event
Description: The median time, in months, from the start of study treatment to an OS event.
Time Frame: Screening, every 4 weeks during treatment (up to 37 weeks), at end of treatment, and every 3 months thereafter
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 5
months | 14.7 [2.5 to NA] — Upper limit of the 95% CI could not be calculated as the follow-up time was too short to observe enough events for complete data estimation.

4. Secondary Outcome: Percentage of Participants Surviving at 12 and 24 Months
Time Frame: Months 12 and 24
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 5
percentage of participants
  12 Months | 60.0 [12.6 to 88.2]
  24 Months | 20.0 [0.8 to 58.2]

5. Primary Outcome: Progression-Free Survival - Time to Event
Description: The median time, in months, from the first study drug treatment to a PFS event.
Time Frame: Screening, every 3 months during treatment (up to 37 weeks), and at end of treatment
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 5
months | 2.5 [0.7 to NA] — Upper limit of the 95 percent (%) confidence interval (CI) could not be calculated as the follow-up time was too short to observe enough events for complete data estimation.

6. Secondary Outcome: Percentage of Participants by Best Overall Response to Treatment
Description: Per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. Complete response (CR) was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal [(short axis less than (<)10 millimeters (mm)]. No new lesions. Partial response (PR) was defined as greater than or equal to (≥)30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. Stable disease (SD) was defined as not qualifying for CR, PR, or progressive disease (PD).
Time Frame: Screening, every 3 months during treatment (up to 37 weeks), and at end of treatment
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 5
percentage of participants
  SD | 20.0
  PD | 80.0
  SD/PD | 100.0

7. Primary Outcome: Percentage of Participants Progression Free at 12 and 24 Months
Time Frame: Months 12 and 24
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 5
percentage of participants
  12 Months | 20.0 [0.8 to 58.2]
  24 Months | 20.0 [0.8 to 58.2]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were recorded from study start to 30 days after the last dose of study drug.
Description: All enrolled participants were included in the safety analysis.
Arm/Group | Trastuzumab Monotherapy
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Monotherapy (N=5)
Pain - stomach (General disorders) | 1
Obstruction - GU (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Monotherapy (N=5)
Pain - extremity, limb (General disorders) | 1
Pain - headache (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Cardiac disorders) | 1
Constitutional symptoms - other (not specified) (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Infection - other (not specified) (Infections and infestations) | 1
Infection with unknown absolute neutrophil count (ANC) (Infections and infestations) | 1
Metabolic/laboratory - other (not specified) (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.